CLINICAL TRIAL: NCT01280500
Title: Accelerating Implementation of Comparative Effectiveness Findings on Clinical and Delivery Systems by Leveraging AHRQ Networks
Brief Title: Title: Comparative Effectiveness of Asthma Interventions Within an AHRQ PBRN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HS10-014
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2018-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Electronic Health Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A - Usual Care Controls (Placebo Comparator): Group A will consist of 20 primary care clinics who are part of the Carolinas Healthcare System network but have not yet adopted the Electronic Medical Record System. These practices do use the same billing databases as the remaining clinics, allowing easy identification of asthma patients and their health services utilization patterns. Data from the billing systems will be used to retrospectively populate a database for these clinics from January 2009 forward.
  Interventions: Other: usual care
- Group B - EMR Control Practices (Active Comparator): There are currently 65 primary care practices within the Carolinas Healthcare System network that have electronic medical record with decision support (EAP)access at baseline. These practices will serve as a second level of control for comparison with the intervention groups. Each of these practices is currently using Cerner PowerChart and at the start of the study and will have access to the asthma decision support tools; an electronically generated Asthma Action Plan (AAP); and a built-in system of population management reports which will be pushed to the practices on an on-going basis to help in patient recall and management. The EAP approach to care has been developed with input from clinicians, hospital administrators, hospital information services personnel, and Cerner consultants.
  Interventions: Behavioral: electronic medical record
- C Integrated Approach to Care (Active Comparator): There are 10 practices within the Carolinas Healthcare System (CHS) network that have already received additional training for improving outcomes for patients with chronic diseases termed the Integrated Approach to Care (IAC). This IAC approach developed by CHS is based on the Chronic Care Model (CCM). The IAC approach includes a heavy emphasis on the use of health information technology that practices receive during the initial EAP rollout.
  Interventions: Other: Integrated Approach to Care
- Group D - Shared Decision Making (SDM) (Active Comparator): This approach has great potential for improved patient outcomes and provides an additional step in the successful implementation of patient self-management. The research team will develop the SDM intervention during the first 6 months of the study. In particular, the Shared decision making (SDM) intervention will be designed to be deployed within the 4 large clinics that care for the majority of the community's underserved and disadvantaged patients. The SDM intervention development will be overseen by the study advisory board and actively recruit providers from within the clinics for feedback about the intervention.
  Interventions: Other: Shared Decision Making
- School Based Care (SBC) (Active Comparator): Activities included: spending individual time with students to assess, treat, and monitor and to educate students in proper asthma management; facilitate access to health care and medicine; and communicate with parents.
  Interventions: Other: school based care

INTERVENTIONS:
Behavioral: electronic medical record — Decision Support, Asthma Action Plans, and Population Management Reporting (EAP)
  Arms: Group B - EMR Control Practices
Other: Integrated Approach to Care — Patients within the IAC group will also receive their own copy of an asthma action plan to allow for some degree of self-management support. In addition, IAC practices receive assistance from a practice coach trained in practice redesign and rapid cycle process improvement.
  Arms: C Integrated Approach to Care
Other: usual care — No EMR
  Arms: Group A - Usual Care Controls
Other: Shared Decision Making — The research team will develop the SDM intervention during the first 6 months of the study. The team will model this intervention on the randomized control trial performed by Dr. Sandra Wilson and colleagues within the Kaiser Permanente Clinics in California and Oregon
  Arms: Group D - Shared Decision Making (SDM)
Other: school based care — the research team will start an electronic data capture system linking school data and the clinical EMR (Cerner Power Chart) that will be implemented over the first year. Flow of data between schools and the hospital system will allow the children who have a regular source of care as well as those without a medical home to be treated with a unified asthma program by the school nurse and the hospital system.
  Arms: School Based Care (SBC)

SUMMARY:
The overall goal is to identify best practices for improving health outcomes for patients with asthma using comparative effectiveness research within an Agency for Healthcare Research and Quality (AHRQ) Practice-Based Research Network (PBRN). This goal will be achieved by completing the following aims: (1) Create a centralized database for comparative effectiveness research on asthma by combining clinical and billing data from one of the largest healthcare systems in the country (Carolinas Healthcare System) with data from the school system, Medicaid, and patient and community-level datasets; (2) Deploy a fully developed integrated approach to asthma management based on the Chronic Care Model; (3) Develop and implement a "shared decision making" approach for asthmatic patients from disadvantaged backgrounds; (4) Implement an electronic data collection system for an existing CDC funded school-based asthma intervention that will allow program evaluation and link school nurses with providers; (5) Evaluate and compare the effectiveness of these three asthma management strategies on: overall healthcare consumption and medical costs; quality of life, school absenteeism and performance; asthma clinical measures; and medication utilization; and (6) Disseminate findings across the state via the statewide PBRN and other network partners. This project has the potential to impact over 30,000 asthma patients across the Carolinas including many patients from disadvantaged backgrounds.

ELIGIBILITY:
Inclusion Criteria:

all with asthma diagnosis

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2011-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Reducing Hospitalizations and Emergency Department Visits | 2011-2013
  Quality goals will be measured by the percentage of patients who reach the goal out of all patients identified with the disease through healthcare system data.

SECONDARY OUTCOMES:
Improving Adherence to Medication | 2011-2013
  Quality goals will be measured by the percentage of patients who reach the goal out of all patients identified with the disease.
Improve Quality of Life | 2011-2013
  Measured via Survey
Reduced School Absenteeism | 2011-2013
  measured with school absenteeism data
Improved Self-Efficacy | 2011-2013
  survey
Improved School Performance | 2011-2013
  measured by yearly end of grade results

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Dulin, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - CMC Elizabeth Family Medicine, Charlotte, North Carolina
  - Department of Family Medicine, Charlotte, North Carolina